CLINICAL TRIAL: NCT00511082
Title: Phase 1 Study of OPB-31121 in Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma or Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 252-07-801-01
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Non-Hodgkin's Lymphoma(NHL); Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Investigational Medicinal Product: OPB-31121 25-mg tablet, 100-mg tablet Dose: OPB-31121 50, 100, 200, 400, 600, 800, and 1000 mg Dosage regimen: ingestion with water after breakfast Treatment period: 4 weeks Mode of Administration: oral administration of OPB-31121 once daily
  Interventions: Drug: OPB-31121

INTERVENTIONS:
Drug: OPB-31121 — 100-mg tablet Dose: OPB-31121 50, 100, 200, 400, 600, 800, and 1000 mg Dosage regimen: ingestion with water after breakfast Treatment period: 4 weeks Mode of Administration: oral administration of OPB-31121 once daily

SUMMARY:
* To investigate the safety and tolerability of OPB-31121 following repeated oral administration of OPB-31121 in patients Non-Hodgkin's Lymphoma(NHL) or Multiple Myeloma(MM)
* To determine the potential dose-limiting toxicities and maximum-tolerated dose in patients treated with OPB-31121
* To determine the pharmacokinetics and anti-tumor efficacy of OPB-31121 in patients

DETAILED DESCRIPTION:
The study is designed as a single-center,open-label,phase 1 dose-escalation study to assess the safety,tolerability,pharmacokinetics, and anti-tumor efficacy of OPB-31121 in patients with relapsed or refractory NHL or MM.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have relapsed or refractory NHL histologically confirmed.
* Relapsed or refractory NHL or MM patients must have experienced treatment failure.
* Chinese patients aged 18 years or older at the time of giving informed consent.
* Performance status score of 0-2 according to the incriteria of he Eastern Cooperative Oncology Group(ECOG)
* Life expectancy of longer than 3 months.
* Patients must have adequate vital organ function.
* Patients are willing to comply with the visit schedules of the hospitalization and outpatient clinic.
* Patients with prior chemotherapy, immunotherapy, cytokines therapy, major surgery, and radiotherapy to the index lesion must have been completed for a minimum period of 4 weeks and recovered from the related toxicity (NCI CTCAE grade 0 or 1) before registration.
* Patients with systemic corticosteroid therapy (>10 mg prednisone or equivalent) must have been completed for a minimum of 1 weeks and recovered from the related toxicity (NCI CTCAE grade 0 or 1) before registration.
* Patients with prior stem cell transplantation must be at least 8 weeks and have recovered from the related toxicity (NCI CTCAE grade 0 or 1) before registration.

Exclusion Criteria:

* Patients are receiving another investigational agent or who have received another investigational agent within 6 months.
* Patients are receiving concurrent chemotherapy, biologic agents, or radiotherapy.
* Patients are receiving concurrent administration of warfarin.
* NHL or MM patients who are candidates for autologous stem cell transplantation are excluded from the study.
* Patients with other primary malignancy except squamous or basal cell skin cancer or cervical cancer in situ.
* Patients with acute lymphoblastic lymphoma/leukaemia, POEMS syndrome or plasma cell leukaemia.
* Lymphoma patients with symptomatic CNS involvement.
* Patients with uncontrolled intercurrent illness.
* Known HIV-positive/AIDS patients.
* Female patients who are pregnant, lactating, or possibly pregnant, or who wish to become pregnant during the study period.
* Patients will not or are unable to use appropriate contraceptive methods during the study period and for at least 6 months after completion of the study
* Patients need to receive any of the following treatments or therapeutic agents during the study period:

  * Anti-cancer drugs other than the study drug
  * Systemic corticosteroid therapy (>10 mg prednisone or equivalent)
  * Radiotherapy as primary therapy
  * Immunotherapy
  * Surgical therapy
  * CYP3A4 and CYP2C9 enzyme inducers or inhibitors,or substrates, and CYP2B6, CYP2C8, and CYP2D6 substrates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 4 weeks

SECONDARY OUTCOMES:
1.Pharmacokinetic Endpoints 2.Efficacy Endpoints & Response Criteria | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenny IK Lei, M.D, Principal Investigator — Department of Clinical Oncology, Prince of Wales Hospital
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No